CLINICAL TRIAL: NCT00420745
Title: Phase IIIb, Double Blind, Randomised, Placebo-Controlled, Multi-Country/Centre, Study to Assess Safety, Reactogenicity & Immunogenicity of 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Pre-Term Infants
Brief Title: To Assess Safety, Reactogenicity & Immunogenicity of 2 Doses of GSK's Oral Human Rotavirus Vaccine in Pre-Term Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 106481
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2009-05-04 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rotarix Group (Experimental): All subjects received 2 oral doses of Rotarix vaccine, 1 dose at Day 0 and 1 dose at Month 1 or 2 depending on the country.
  Interventions: Biological: Rotarix™
- Placebo Group (Placebo Comparator): All subjects received 2 oral doses of placebo, 1 dose at Day 0 and 1 dose at Month 1 or 2 depending on the country.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix™ — Two-dose oral vaccination.
  Arms: Rotarix Group
Biological: Placebo — Two-dose oral administration
  Arms: Placebo Group

SUMMARY:
This study is planned to evaluate the safety (in terms of occurrence of any serious adverse events), reactogenicity (any side effects) and immunogenicity (ability of the vaccine to develop antibodies that fight infection) of the HRV vaccine when used in pre-term infants aged between 6 and 14 weeks at the time of the first dose in Portugal, France and Poland and in pre-term infants aged between 6 and 12 weeks at the time of first dose in Spain. The study will be performed in four European countries (France, Poland, Spain, and Portugal). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This is a Phase 3b study.

Each study group is further stratified into two sub-groups depending on the gestational age at birth of the subject:

* Stratum I: very pre-term infants, born after a gestational period of 27-30 weeks (189-216 days) (20% of enrolment).
* Stratum II: mild pre-term infants born after a gestational period of 31-36 weeks (217-258 days) (80% of enrolment).

The study will be conducted in a double-blind manner with respect to the HRV vaccine and placebo. The study will not be blinded with respect to the type of concomitantly administered routine infant vaccination.

In accordance with the local National Plan of Immunisation schedule in each of the respective participating countries, GSK Biologicals' Infanrix Hexa™ (DTPa-HBV-IPV/Hib), Infanrix Quinta™ (DTPa-IPV-Hib), Infanrix™+IPV+Hib (DTPa+IPV+Hib) and/or Engerix-B™ (HBV) will be co-administered (at a maximum interval of two days from each other) with each HRV vaccine or placebo dose.

Hepatitis B and Bacille Calmette-Guérin vaccines (BCG) at birth are allowed if included in the local National Plan of Immunisation schedule in participating countries.

At the discretion of the investigator the following vaccines may be administered during each subject's study participation:

* Vaccine against Streptococcus pneumoniae (Prevenar®) in France and Spain (concomitantly with HRV vaccine/Placebo).
* Vaccine against Neisseria meningitidis (Neis Vacc C®) is allowed if there is at least 14-days interval with respect to the administration of the HRV vaccine/Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Healthy male or female infant between, and including, 6 and 14 weeks (42 - 104 days) of age at the time of first study vaccination in Portugal, France and Poland. A male or female infant between, and including, 6 and 12 weeks of age at the time of first study vaccination in Spain.
* Medically stable pre-term infants, born within a gestational period of 27 -36 weeks.
* Written informed consent obtained from the parent or guardian of the subject.
* Planned to be discharged from hospital's neonatal stay on or before the day of the first HRV vaccine/Placebo administration.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the HRV vaccine within 30 days preceding the first dose of HRV vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccines not foreseen by the study protocol from birth till study end.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any clinically significant history of chronic gastrointestinal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness (subjects with severe broncho-pulmonary dysplasia requiring persistent oxygen-therapy will be excluded).
* History of any neurologic disorders or seizures. Grade I and II intra-ventricular bleeding are allowed.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins, and/or any blood products within one month (30 days) preceding the first dose of study vaccines or planned administration during the study period. Monoclonal anti-RSV therapy/prophylaxis and recombinant erythropoietin are allowed.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1009 (Actual)
Dates: Start 2007-01-25; Primary Completion 2008-03-01 (Actual); Study Completion 2008-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- France (8):
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
- Poland (8):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Mielec
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw
- Portugal (3):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Spain (9):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Fuenlabrada (Madrid)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Omenaca F, Sarlangue J, Szenborn L, Nogueira M, Suryakiran PV, Smolenov IV, Han HH; ROTA-054 Study Group. Safety, reactogenicity and immunogenicity of the human rotavirus vaccine in preterm European Infants: a randomized phase IIIb study. Pediatr Infect Dis J. 2012 May;31(5):487-93. doi: 10.1097/INF.0b013e3182490a2c. PMID 22228231
- [Background] Omenaca F et al. Immunogenicity of a rotavirus vaccine (RIX4414) in European pre-term infants with different gestational age. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Omenaca F et al. Safety, Reactogenicity and Immunogenicity of RIX4414 Live Attenuated Human Rotavirus Vaccine in Pre-Term Infants. Abstract presented at the ICAAC/IDSA Joint Meeting, Washington DC, US, 25-28 October 2008.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106481 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 670 | 339
Completed | 655 | 333
Not Completed | 15 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 10 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Recurrent pneumonia & bronchitis | 0 | 1
Not completed — Age limit exceeded for Dose 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 670 | 339 | 1009
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.5 (1.77) | 8.5 (1.78) | 8.5 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 167 | 494
  Male | 343 | 172 | 515

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From Day 0 up to 1 month after Dose 2 of Rotarix vaccine/Placebo
Population: The analyses were performed on the Total Vaccinated Cohort that included all the subjects with at least one study vaccine or placebo administration documented.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 670 | 339
subjects | 34 | 23

2. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs), According to Medical Dictionary for Regulatory Activities (MedDRA) Classification.
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 31 days after any Rotarix vaccine/Placebo dose.
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 670 | 339
subjects | 196 | 138

3. Secondary Outcome: Number of Subjects for Whom Each Type of Solicited Symptom Was Reported.
Description: Solicited symptoms included Diarrhea (3 or more looser than normal stools/day), Fever (axillary temperature ≥ 37.5 degrees Celsius (°C)), Irritability, Loss of appetite, and Vomiting
Time Frame: Within 15 days after each Rotarix vaccine/Placebo dose.
Population: The analyses were performed on the Total vaccinated cohort for the safety and the immunogenicity subset that included all subjects with at least one study vaccine or placebo administered and for whom solicited symptoms were collected.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 203 | 100
subjects
  Diarrhea | 9 | 5
  Fever | 54 | 29
  Irritability | 133 | 66
  Loss of appetite | 81 | 45
  Vomiting | 52 | 27

4. Secondary Outcome: Number of Subjects for Whom Presence of Rotavirus (RV) Gastroenteritis (GE) Was Detected in Stools.
Description: Gastroenteritis (GE): diarrhoea with or without vomiting. Rotavirus (RV) GE: A GE episode was a RV GE if a stool sample taken during or not later than 7 days after the episode was RV positive by Enzyme Linked Immunosorbent Assay.
Time Frame: From Dose 1 up to 1 month after Dose 2 of Rotarix vaccine/Placebo
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 670 | 339
subjects | 3 | 2

5. Secondary Outcome: Seroconversion to Anti-rotavirus Immunoglobulin A (IgA) Antibody.
Description: Number of subjects with anti-rotavirus IgA antibody concentration ≥ 20 Units/milliliter (U/mL).
Time Frame: At Visit 3, 1 month after Dose 2 of Rotarix vaccine/Placebo
Population: The analyses were performed on the According-to-Protocol immunogenicity cohort that included all subjects with at least one study vaccine or placebo administered, for whom immunogenicity data were collected and available and who complied with the inclusion criteria defined in the protocol.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 147 | 81
subjects | 126 | 13

6. Secondary Outcome: Serum Anti-Rotavirus IgA Antibody Concentration.
Description: Anti-rotavirus IgA antibody concentrations are given as geometric mean concentrations (GMC) with 95% Confidence Intervals, calculated on all subjects.
Time Frame: At Visit 3, 1 month after Dose 2 of Rotarix vaccine/Placebo
Population: The analyses were performed on the According-to-Protocol immunogenicity cohort. The anti-rotavirus IgA antibody GMC for Placebo Group was below the assay cut-off (<20 U/mL), so could not be computed.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 147 | 0
U/mL | 202.2 [153.1 to 267.1] |

ADVERSE EVENTS:
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 34 | 23
Other Adverse Events (participants affected / at risk) | 199/670 | 110/339
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Rotarix Group | Placebo Group
Anaemia (Blood and lymphatic system disorders) | 0/670 | 2/339
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1/670 | 0/339
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1/670 | 0/339
Bronchiolitis (Infections and infestations) | 3/670 | 4/339
Bronchitis (Infections and infestations) | 4/670 | 2/339
Bronchopneumonia (Infections and infestations) | 4/670 | 1/339
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1/670 | 0/339
Cough (Respiratory, thoracic and mediastinal disorders) | 0/670 | 1/339
Dacryocystitis (Infections and infestations) | 1/670 | 0/339
Dehydration (Metabolism and nutrition disorders) | 1/670 | 0/339
Diarrhoea (Gastrointestinal disorders) | 2/670 | 0/339
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0/670 | 1/339
Dyspepsia (Gastrointestinal disorders) | 0/670 | 2/339
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/670 | 1/339
Gastritis (Gastrointestinal disorders) | 1/670 | 0/339
Gastroenteritis (Gastrointestinal disorders) | 6/670 | 1/339
Gastroenteritis adenovirus (Infections and infestations) | 0/670 | 1/339
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/670 | 1/339
Gastroenteritis rotavirus (Infections and infestations) | 0/670 | 1/339
Hyperkalaemia (Metabolism and nutrition disorders) | 0/670 | 1/339
Hypernatraemia (Metabolism and nutrition disorders) | 1/670 | 0/339
Inguinal hernia (Gastrointestinal disorders) | 0/670 | 2/339
Nephrolithiasis (Renal and urinary disorders) | 0/670 | 1/339
Otitis media acute (Infections and infestations) | 0/670 | 1/339
Periorbital cellulitis (Infections and infestations) | 1/670 | 0/339
Pertussis (Infections and infestations) | 1/670 | 0/339
Pneumonia (Infections and infestations) | 4/670 | 2/339
Pneumonia bacterial (Infections and infestations) | 0/670 | 1/339
Pyelonephritis acute (Infections and infestations) | 2/670 | 0/339
Pyrexia (General disorders) | 4/670 | 3/339
Rectal haemorrhage (Gastrointestinal disorders) | 1/670 | 0/339
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2/670 | 3/339
Respiratory tract infection (Infections and infestations) | 0/670 | 1/339
Sepsis (Infections and infestations) | 1/670 | 0/339
Urinary tract infection (Infections and infestations) | 1/670 | 0/339
OTHER ADVERSE EVENTS (reported when occurring in more than 1.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=670) | Placebo Group (N=339)
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Fever (General disorders) | 54 | 29
Irritability (General disorders) | 133 | 66
Loss of appetite (Metabolism and nutrition disorders) | 81 | 45
Vomiting (Gastrointestinal disorders) | 52 | 27
Pyrexia (General disorders) | 28 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.